CLINICAL TRIAL: NCT05041114
Title: Stentrode With Thought-controlled Digital Switch: An Early Feasibility Study of the Safety of an Endovascular Motor Neuroprosthesis in Participants With Severe Upper Limb Impairment.
Brief Title: SWITCH II Early Feasibility Study: Implantable BCI to Control a Digital Device for People With Paralysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study moved to U.S.
Sponsor: Synchron Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: Synchron, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-01-02
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Neurologic Disorder; Paralysis; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Spinal Cord Injury; Stroke, Lacunar; Stroke, Brainstem; Upper Limb Injury; Spinal Muscular Atrophy
MeSH Terms: conditions — Nervous System Diseases; Paralysis; Stroke; Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Spinal Cord Injuries; Stroke, Lacunar; Brain Stem Infarctions; Arm Injuries; Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Other): Implantation of motor neuroprosthesis medical device.
  Interventions: Device: Motor Neuroprosthesis

INTERVENTIONS:
Device: Motor Neuroprosthesis — Type of implantable brain computer interface

SUMMARY:
The Synchron Motor Neuroprosthesis (MNP) is intended to be used in subjects with severe motor impairment, unresponsive to medical or rehabilitative therapy and a persistent functioning motor cortex. The purpose of this research is to evaluate safety and feasibility.

The MNP is a type of implantable brain computer interface which bypasses dysfunctional motor neurons. The device is designed to restore the transmission of neural signal from the cerebral cortex utilized for neuromuscular control of digital devices, resulting in a successful execution of non-mechanical digital commands.

ELIGIBILITY:
Inclusion Criteria:

1. Severe motor impairment
2. Able to give consent
3. Appropriate candidate for neurointerventional procedure
4. Able and willing to access all clinical testing and not impeded by geographical location
5. Proficient in English
6. Have a study partner

Exclusion Criteria:

1. Active condition resulting in immunosuppression
2. Unsuitable for general anaesthetic
3. Anaphylactic allergy to contrast media
4. Allergy to nickel
5. History of pulmonary embolism
6. History of recent deep vein thrombosis
7. Psychiatric or psychological disorder
8. No study partner or caregiver
9. Unable to provide evidence of COVID vaccination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | 12 months post implant

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Sydney Local Health District, Sydney, New South Wales
  - Metro North Health, Brisbane, Queensland
  - Melbourne Health, Melbourne, Victoria